CLINICAL TRIAL: NCT05064488
Title: A Phase I, Open-Label, Two-Part Study of the Effect of Multiple-Dose Evobrutinib on Transporter Substrates Digoxin, Metformin, Rosuvastatin, and Sumatriptan Pharmacokinetics in Healthy Participants
Brief Title: Drug-Drug Interaction Study of Evobrutinib and Transporter Substrates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS200527_0078; 2021-001923-42 (EudraCT Number)
Record Dates: First submitted 2021-09-23; First posted 2021-10-01 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Clinical Pharmacology; Drug interaction; Evobrutinib; Digoxin; Metformin; Rosuvastatin; Sumatriptan
MeSH Terms: interventions — evobrutinib; Digoxin; Metformin; Rosuvastatin Calcium; Sumatriptan

STUDY DESIGN:
Intervention Model Description: single-sequence study (each part)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1: Cocktail (Day 1) (Experimental): Participants received single oral dose of Cocktail (digoxin 0.25 mg tablet, metformin 10 mg solution, rosuvastatin 10 mg tablet) on Day 1 in Part 1 under fed conditions.
  Interventions: Drug: Digoxin (0.25mg); Drug: Metformin (10mg); Drug: Rosuvastatin (10mg)
- Part 1: Evobrutinib (Days 4 to 12) (Experimental): Participants received Evobrutinib film-coated tablets, at a dose of 45 mg, orally, twice a day on Days 4 to 12 in Part 1 under fed conditions.
  Interventions: Drug: Evobrutinib (45mg)
- Part 1: Evobrutinib + Cocktail (Day 10) (Experimental): Participants received Evobrutinib film-coated tablets, at a dose of 45 mg, orally, twice a day and cocktail (digoxin 0.25 mg tablet, metformin 10 mg solution, rosuvastatin 10 mg tablet) on Day 10 in Part 1 under fed conditions.
  Interventions: Drug: Evobrutinib (45mg); Drug: Digoxin (0.25mg); Drug: Metformin (10mg); Drug: Rosuvastatin (10mg)
- Part 2: Sumatriptan (Day 1) (Experimental): Participants received single oral dose of Sumatriptan 25 mg tablet on Day 1 in Part 2 under fed conditions.
  Interventions: Drug: Sumatriptan (25mg)
- Part 2: Evobrutinib (Days 2 to 8) (Experimental): Participants received Evobrutinib film-coated tablets, at a dose of 45 mg, orally, twice a day on Days 2 to 8 in Part 2 under fed conditions.
  Interventions: Drug: Evobrutinib (45mg)
- Part 2: Evobrutinib + Sumatriptan (Day 8) (Experimental): Participants received Evobrutinib film-coated tablets, at a dose of 45 mg, orally, twice a day and single oral dose of Sumatriptan 25 mg tablet on Day 8 in Part 2 under fed conditions.
  Interventions: Drug: Evobrutinib (45mg); Drug: Sumatriptan (25mg)

INTERVENTIONS:
Drug: Evobrutinib (45mg) — Participants received film-coated Evobrutinib tablet at a dose of 45 milligrams (mg), orally twice daily on Days 4 to 12 in Part 1 and Days 2 to 8 in Part 2 under fed conditions.
  Other Names: M2951
  Arms: Part 1: Evobrutinib (Days 4 to 12); Part 1: Evobrutinib + Cocktail (Day 10); Part 2: Evobrutinib (Days 2 to 8); Part 2: Evobrutinib + Sumatriptan (Day 8)
Drug: Digoxin (0.25mg) — Participants received single oral dose of digoxin tablet (0.25 mg) on Day 1 and Day 10 in Part 1 under fed conditions.
  Arms: Part 1: Cocktail (Day 1); Part 1: Evobrutinib + Cocktail (Day 10)
Drug: Metformin (10mg) — Participants received single oral dose of metformin 10 mg solution on Day 1 and Day 10 in Part 1 under fed conditions.
  Arms: Part 1: Cocktail (Day 1); Part 1: Evobrutinib + Cocktail (Day 10)
Drug: Rosuvastatin (10mg) — Participants received single oral dose of rosuvastatin tablet (10 mg) on Day 1 and Day 10 in Part 1 under fed conditions.
  Arms: Part 1: Cocktail (Day 1); Part 1: Evobrutinib + Cocktail (Day 10)
Drug: Sumatriptan (25mg) — Participants received single dose of sumatriptan tablet (25 mg) on Day 1 and Day 8 in Part 2 under fed conditions.
  Arms: Part 2: Evobrutinib + Sumatriptan (Day 8); Part 2: Sumatriptan (Day 1)

SUMMARY:
This study consisted of 2 parts: Part 1 and 2. The purpose of this study was to evaluate the pharmacokinetic, safety and tolerability of multiple doses of evobrutinib on single doses of digoxin, metformin and rosuvastatin in Part-1 and sumatriptan in Part-2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants were overtly healthy as determined by medical evaluation, including no clinically significant abnormality identified on physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion
* Participants had a body weight within 50.0 and 100.0 kilograms [kg] (inclusive) and body mass index within the range of 19.0 and 30.0 kilograms per square meter [kg/m^2] (inclusive)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders, as determined by medical evaluation
* Individuals with diagnosis of hemochromatosis, Wilson´s disease, alpha 1 antitrypsin deficiency, or any other chronic liver disease including Gilbert's disease were excluded from the study
* Prior history of cholecystectomy or splenectomy, and any clinically relevant surgery within 6 months prior to Screening
* History of any malignancy
* History of chronic or recurrent acute infection or any bacterial, viral, parasitic or fungal infections within 30 days prior to Screening and at any time between Screening and admission, or hospitalization due to infection within 6 months prior to Screening
* History of shingles within 12 months prior to Screening
* History of drug hypersensitivity, ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients; history of serious allergic reactions leading to hospitalization or any other hypersensitivity reaction in general, which may affect the safety of the participant and/or outcome of the study per the Investigator's discretion
* History of alcoholism or drug abuse within 2 years prior to Screening, or positive for drugs of abuse, nicotine/cotinine or alcohol by the laboratory assays conducted during Screening and Day -1
* History of residential exposure to tuberculosis, or a positive QuantiFERON® test within 4 weeks prior to or at the time of Screening
* Administration of live vaccines or live-attenuated virus vaccines within 3 months prior to Screening
* Moderate or strong inhibitors or inducers of Cytochrome P450, family 3, subfamily A (CYP3A4/5) within 4 weeks prior to the first administration of study intervention
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0078
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 40 healthy participants were enrolled in two parts single-sequences: Part 1 (Evobrutinib and Cocktail [digoxin, metformin, and rosuvastatin] as transporter substrates) and Part 2 (Evobrutinib and Sumatriptan as transporter substrate) with each part consists of 20 participants.
Groups:
- Part 1: All Participants: Participants received single oral dose of Cocktail (digoxin 0.25 milligrams [mg] tablet, metformin 10 mg solution, rosuvastatin 10 mg tablet) on Days 1 and 10; Evobrutinib film-coated tablets at a dose of 45 mg, orally, twice daily on Days 4 to 12 in Part 1 under fed conditions.
- Part 2: All Participants: Participants received single oral dose of Sumatriptan tablet 25 mg on Days 1 and 8; Evobrutinib film-coated tablets at a dose of 45 mg, orally, twice daily on Days 2 to 8 in Part 2 under fed conditions.
Period: Overall Study
Arm/Group | Part 1: All Participants | Part 2: All Participants
Started | 20 | 20
Part 1: Cocktail (Day 1) | 20 (Participant dropped out on Day 11 after the evobrutinib morning dose and 1 participant dropped out on Day 6 after the evobrutinib morning dose.) | 0
Part 1: Evobrutinib + Cocktail (Day 10) | 19 (Evobrutinib administration in 1 participant was stopped on Day 6 after the morning dose and the participant did not receive the evobrutinib + cocktail on Day 10.) | 0
Part 2: Sumatriptan (Day 1) | 0 | 20
Part 2: Evobrutinib (Days 2 to 8) | 0 | 20
Part 2: Evobrutinib + Sumatriptan (Day 8) | 0 | 20
Part 1: Evobrutinib (Days 4 to 12) | 20 (1 Participant dropped out on Day 11 after the evobrutinib morning dose and 1 participant dropped out on Day 6 after the evobrutinib morning dose.) | 0
Completed | 18 | 20
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: All Participants | Part 2: All Participants | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 9 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Digoxin
Description: The AUC from time zero (= dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from lambda z determination: AUC0-inf= AUC0-tlast + Clast pred/lambda z, where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down); Clast pred was defined as the predicted concentration at the last sampling time, calculated from the log-linear regression line for lambda z determination and Lambda z was the apparent terminal rate constant. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on digoxin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: Pharmacokinetic (PK) population included all participants who have completed the study without any relevant protocol deviations and factors likely to affect the comparability of PK results, with adequate study intervention compliance.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter (h*ng/mL)
Groups:
- Part 1: Cocktail: Participants received single oral dose of Cocktail (digoxin 0.25 mg tablet, metformin 10 mg solution, rosuvastatin 10 mg tablet) on Day 1 in Part 1 under fed conditions.
- Part 1: Evobrutinib + Cocktail: Participants received Evobrutinib film-coated tablets, at a dose of 45 mg, orally, twice a day and cocktail (digoxin 0.25 mg tablet, metformin 10 mg solution, rosuvastatin 10 mg tablet) on Day 10 in Part 1 under fed conditions.
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
Hour*nanogram per milliliter (h*ng/mL) | 15.8 (21.5) | 18.7 (23.7)
Statistical Analysis 1: Comparison: Part 1: Cocktail vs Part 1: Evobrutinib + Cocktail; Treatment differences on the log scale of transporter substrates with evobrutinib vs substrates alone; Test type: Other — A general linear model with a fixed effect for treatment and a random effect for participant was applied to log-transformed PK parameters AUC0-inf based on the PK analysis set to assess the effect of multiple doses of evobrutinib on the PK of the transporter substrates digoxin; Ratio = 118.49, 90% CI 2-sided [111.89 to 125.47]

2. Primary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Metformin
Description: The AUC from time zero (= dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from lambda z determination: AUC0-inf= AUC0-tlast + Clast pred/lambda z, where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down); Clast pred was defined as the predicted concentration at the last sampling time, calculated from the log-linear regression line for lambda z determination and Lambda z was the apparent terminal rate constant. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on metformin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: PK population included all participants who have completed the study without any relevant protocol deviations and factors likely to affect the comparability of PK results, with adequate study intervention compliance.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
h*ng/mL | 20.2 (23.3) | 42.2 (77.1)
Statistical Analysis 1: Comparison: Part 1: Cocktail vs Part 1: Evobrutinib + Cocktail; Treatment differences on the log scale of transporter substrates with evobrutinib vs substrates alone; Test type: Other — A general linear model with a fixed effect for treatment and a random effect for participant was applied to log-transformed PK parameters AUC0-inf based on the PK analysis set to assess the effect of multiple doses of evobrutinib on the PK of the transporter substrates metformin; Ratio = 208.95, 90% CI 2-sided [155.48 to 280.82]

3. Primary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Rosuvastatin
Description: The AUC from time zero (= dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from lambda z determination: AUC0-inf= AUC0-tlast + Clast pred/lambda z, where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down); Clast pred was defined as the predicted concentration at the last sampling time, calculated from the log-linear regression line for lambda z determination and Lambda z was the apparent terminal rate constant. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on rosuvastatin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: PK population included all participants who have completed the study without any relevant protocol deviations and factors likely to affect the comparability of PK results, with adequate study intervention compliance. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 11 | 11
h*ng/mL | 34.6 (64.3) | 34.3 (74.7)
Statistical Analysis 1: Comparison: Part 1: Cocktail vs Part 1: Evobrutinib + Cocktail; Treatment differences on the log scale of transporter substrates with evobrutinib vs substrates alone; Test type: Other — A general linear model with a fixed effect for treatment and a random effect for participant was applied to log-transformed PK parameters AUC0-inf based on the PK analysis set to assess the effect of multiple doses of evobrutinib on the PK of the transporter substrates rosuvastatin; Ratio = 99.05, 90% CI 2-sided [80.49 to 121.89]

4. Primary Outcome: Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Sumatriptan
Description: The AUC from time zero (= dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from lambda z determination: AUC0-inf= AUC0-tlast + Clast pred/lambda z, where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down); Clast pred was defined as the predicted concentration at the last sampling time, calculated from the log-linear regression line for lambda z determination and Lambda z was the apparent terminal rate constant. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on sumatriptan in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Part 2: Sumatriptan: Participants received single oral dose of Sumatriptan 25 mg tablet on Day 1 in Part 2 under fed conditions.
- Part 2: Evobrutinib + Sumatriptan: Participants received Evobrutinib film-coated tablets, at a dose of 45 mg, orally, twice a day and single oral dose of Sumatriptan 25 mg tablet on Day 8 in Part 2 under fed conditions.
Arm/Group | Part 2: Sumatriptan | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 19 | 19
h*ng/mL | 52.5 (43.7) | 46.9 (41.0)
Statistical Analysis 1: Comparison: Part 2: Sumatriptan vs Part 2: Evobrutinib + Sumatriptan; Treatment differences on the log scale of transporter substrates with evobrutinib vs substrates alone; Test type: Other — A general linear model with a fixed effect for treatment and a random effect for participant was applied to log-transformed PK parameters AUC0-inf based on the PK analysis set to assess the effect of multiple doses of evobrutinib on the PK of the transporter substrates sumatriptan; Ratio = 89.35, 90% CI [82.70 to 96.54]

5. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Digoxin
Description: Cmax was obtained directly from the concentration versus time curve. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on digoxin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
Nanogram per milliliter (ng/mL) | 1.15 (31.7) | 1.15 (34.8)
Statistical Analysis 1: Comparison: Part 1: Cocktail vs Part 1: Evobrutinib + Cocktail; Treatment differences on the log scale of transporter substrates with evobrutinib vs substrates alone; Test type: Other — A general linear model with a fixed effect for treatment and a random effect for participant was applied to log-transformed PK parameters Cmax based on the PK analysis set to assess the effect of multiple doses of evobrutinib on the PK of the transporter substrates digoxin; Ratio = 100.64, 90% CI 2-sided [85.99 to 117.79]

6. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Metformin
Description: Cmax was obtained directly from the concentration versus time curve. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on metformin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
ng/mL | 3.24 (23.1) | 6.58 (76.5)
Statistical Analysis 1: Comparison: Part 1: Cocktail vs Part 1: Evobrutinib + Cocktail; Treatment differences on the log scale of transporter substrates with evobrutinib vs substrates alone; Test type: Other — A general linear model with a fixed effect for treatment and a random effect for participant was applied to log-transformed PK parameters Cmax based on the PK analysis set to assess the effect of multiple doses of evobrutinib on the PK of the transporter substrates metformin; Ratio = 203.08, 90% CI 2-sided [152.93 to 269.68]

7. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Rosuvastatin
Description: Cmax was obtained directly from the concentration versus time curve. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on rosuvastatin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 11 | 11
ng/mL | 2.35 (60.3) | 2.16 (66.5)
Statistical Analysis 1: Comparison: Part 1: Cocktail vs Part 1: Evobrutinib + Cocktail; Treatment differences on the log scale of transporter substrates with evobrutinib vs substrates alone; Test type: Other — A general linear model with a fixed effect for treatment and a random effect for participant was applied to log-transformed PK parameters Cmax based on the PK analysis set to assess the effect of multiple doses of evobrutinib on the PK of the transporter substrates rosuvastatin; Ratio = 91.74, 90% CI 2-sided [76.98 to 109.33]

8. Primary Outcome: Part 2: Maximum Observed Plasma Concentration (Cmax) of Sumatriptan
Description: Cmax was obtained directly from the concentration versus time curve. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on sumatriptan in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Sumatriptan | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 19 | 19
ng/mL | 13.4 (39.7) | 10.9 (38.6)
Statistical Analysis 1: Comparison: Part 2: Sumatriptan vs Part 2: Evobrutinib + Sumatriptan; Treatment differences on the log scale of transporter substrates with evobrutinib vs substrates alone; Test type: Other — A general linear model with a fixed effect for treatment and a random effect for participant was applied to log-transformed PK parameters Cmax based on the PK analysis set to assess the effect of multiple doses of evobrutinib on the PK of the transporter substrates sumatriptan; Ratio = 81.02, 90% CI 2-sided [74.23 to 88.42]

9. Secondary Outcome: Part 1 and Part 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether considered related to the study intervention or not. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE: AE with onset after start of treatment or with onset date before the treatment start date but worsening after the treatment start date. TEAEs included both serious and non-serious TEAEs.
Time Frame: Part 1: Cocktail Alone - Day 1 to Day 3; Evobrutinib Alone - Day 4 to Day 9; Evobrutinib + Cocktail - Day 10 to Day 12; Part 2: Sumatriptan Alone - Day 1; Evobrutinib Alone - Day 2 to Day 7; Evobrutinib + Sumatriptan - Day 8
Population: The safety analysis set (SAF) included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Evobrutinib: Participants received Evobrutinib film-coated tablets, at a dose of 45 mg, orally, twice a day on Days 4 to 12 in Part 1 under fed conditions.
- Part 2: Evobrutinib: Participants received Evobrutinib film-coated tablets, at a dose of 45 mg, orally, twice a day on Days 2 to 8 in Part 2 under fed conditions.
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib | Part 1: Evobrutinib + Cocktail | Part 2: Sumatriptan | Part 2: Evobrutinib | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 20 | 20 | 19 | 20 | 20 | 20
Participants
  Participants with TEAEs | 7 | 9 | 6 | 6 | 10 | 8
  Participants with Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Part 1 and Part 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs) by Severity
Description: Severity of TEAEs were graded using Qualitative Toxicity Scale, as follows: Mild: Participant is aware of the event or symptom, but the event or symptom is easily tolerated; Moderate: Participant experiences sufficient discomfort to interfere with or reduce his or her usual level of activity; Severe: Significant impairment of functioning: the participant is unable to carry out his or her usual activities. Number of participants with TEAEs by severity were reported.
Time Frame: as for outcome 9
Population: The SAF included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib | Part 1: Evobrutinib + Cocktail | Part 2: Sumatriptan | Part 2: Evobrutinib | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 20 | 20 | 19 | 20 | 20 | 20
Participants
  Mild TEAEs | 5 | 9 | 6 | 4 | 10 | 7
  Moderate TEAEs | 3 | 1 | 1 | 2 | 0 | 2
  Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Part 1 and Part 2: Number of Participants With Clinically Relevant Changes From Baseline in Laboratory Parameters
Description: Laboratory investigation included hematology, biochemistry and urinalysis. Clinical meaningful changes were determined by the investigator. The number of participants with clinically relevant changes from baseline in laboratory parameters were reported.
Time Frame: as for outcome 9
Population: The SAF included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib | Part 1: Evobrutinib + Cocktail | Part 2: Sumatriptan | Part 2: Evobrutinib | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 20 | 20 | 19 | 20 | 20 | 20
Participants | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Part 1 and Part 2: Number of Participants With Clinically Relevant Changes From Baseline in Vital Signs
Description: Vital signs included body temperature, systolic and diastolic blood pressure and pulse rate. Clinical relevance was determined by the investigator. The number of participants with clinically relevant changes from baseline in vital signs were reported.
Time Frame: as for outcome 9
Population: The SAF included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib | Part 1: Evobrutinib + Cocktail | Part 2: Sumatriptan | Part 2: Evobrutinib | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 20 | 20 | 19 | 20 | 20 | 20
Participants | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Part 1 and Part 2: Number of Participants With Clinically Relevant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Findings
Description: 12-lead ECG recordings included rhythm, heart rate (as measured by RR interval), PR interval, QRS duration and QT interval. The corrected QT interval (QTcF) was calculated using Fridericia's formula. 12-lead ECG recordings were obtained after the participants have rested for at least 10 minutes in semisupine position. Clinical relevance was determined by the investigator. The number of participants with clinically relevant changes from baseline in 12-Lead ECG findings were reported.
Time Frame: as for outcome 9
Population: The SAF included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib | Part 1: Evobrutinib + Cocktail | Part 2: Sumatriptan | Part 2: Evobrutinib | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 20 | 20 | 19 | 20 | 20 | 20
Participants | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Digoxin
Description: Tmax was the time to reach the maximum observed concentration collected during a dosing interval. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on digoxin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
Hours | 1.50 [0.333 to 2.00] | 2.00 [0.667 to 4.00]

15. Secondary Outcome: Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Metformin
Description: Tmax was the time to reach the maximum observed concentration collected during a dosing interval. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on metformin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
Hours | 3.00 [3.00 to 4.02] | 4.00 [2.00 to 4.02]

16. Secondary Outcome: Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Rosuvastatin
Description: Tmax was the time to reach the maximum observed concentration collected during a dosing interval. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on rosuvastatin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 11 | 11
Hours | 4.00 [1.50 to 8.00] | 4.00 [1.50 to 6.02]

17. Secondary Outcome: Part 2: Time to Reach Maximum Plasma Concentration (Tmax) of Sumatriptan
Description: Tmax was the time to reach the maximum observed concentration collected during a dosing interval. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on sumatriptan in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 8
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Sumatriptan | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 19 | 19
Hours | 2.00 [1.50 to 3.05] | 2.00 [1.50 to 4.00]

18. Secondary Outcome: Part 1: Apparent Terminal Half-Life (t1/2) of Digoxin
Description: T1/2 was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half. T1/2 was calculated by natural log 2 divided by Lambda z. Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on digoxin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
Hours | 31.0 [24.1 to 67.9] | 46.9 [24.6 to 69.4]

19. Secondary Outcome: Part 1: Apparent Terminal Half-Life (t1/2) of Metformin
Description: T1/2 was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half. T1/2 was calculated by natural log 2 divided by Lambda z. Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method. The transporter cocktail included digoxin, metformin, and rosuvastatin.
  As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on metformin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
Hours | 3.02 [2.52 to 5.24] | 3.50 [2.23 to 13.8]

20. Secondary Outcome: Part 1: Apparent Terminal Half-Life (t1/2) of Rosuvastatin
Description: T1/2 was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half. T1/2 was calculated by natural log 2 divided by Lambda z. Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method. The transporter cocktail included digoxin, metformin, and rosuvastatin.
  As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on rosuvastatin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 11 | 11
Hours | 15.5 [12.5 to 29.1] | 15.5 [9.60 to 19.0]

21. Secondary Outcome: Part 2: Apparent Terminal Half-Life (t1/2) of Sumatriptan
Description: T1/2 was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half. T1/2 was calculated by natural log 2 divided by Lambda z. Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on sumatriptan in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 8
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Sumatriptan | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 19 | 19
Hours | 3.16 [1.45 to 8.73] | 3.56 [1.60 to 8.77]

22. Secondary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Sampling Time (AUC0-tlast) of Digoxin
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification was calculated using the mixed log-linear trapezoidal rule (linear up, log down). The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on digoxin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
h*ng/mL | 12.1 (21.3) | 12.9 (23.4)
Statistical Analysis 1: Comparison: Part 1: Cocktail vs Part 1: Evobrutinib + Cocktail; Test type: Other; Ratio = 106.83, 90% CI 2-sided [102.11 to 111.76]

23. Secondary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Sampling Time (AUC0-tlast) of Metformin
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification was calculated using the mixed log-linear trapezoidal rule (linear up, log down). The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on metformin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
h*ng/mL | 19.5 (23.7) | 41.3 (79.2)
Statistical Analysis 1: Comparison: Part 1: Cocktail vs Part 1: Evobrutinib + Cocktail; Test type: Other; Ratio = 211.42, 90% CI 2-sided [156.34 to 285.91]

24. Secondary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Sampling Time (AUC0-tlast) of Rosuvastatin
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification was calculated using the mixed log-linear trapezoidal rule (linear up, log down). The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on rosuvastatin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 11 | 11
h*ng/mL | 31.0 (65.0) | 30.9 (80.6)
Statistical Analysis 1: Comparison: Part 1: Cocktail vs Part 1: Evobrutinib + Cocktail; Test type: Other; Ratio = 99.57, 90% CI 2-sided [79.69 to 124.42]

25. Secondary Outcome: Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Sampling Time (AUC0-tlast) of Sumatriptan
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification was calculated using the mixed log-linear trapezoidal rule (linear up, log down). As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on sumatriptan in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2: Sumatriptan | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 19 | 19
h*ng/mL | 51.2 (44.4) | 45.5 (41.7)
Statistical Analysis 1: Comparison: Part 2: Sumatriptan vs Part 2: Evobrutinib + Sumatriptan; Test type: Other; Ratio = 88.83, 90% CI 2-sided [82.04 to 96.19]

26. Secondary Outcome: Part 1: Apparent Total Body Clearance From Plasma (CL/F) of Digoxin
Description: CL/f was calculated as Dose/AUC0-inf, where AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. AUC0-inf was calculated as AUC0-tlast + Clast pred/Lambda Z, where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification; Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the lower limit of quantification (LLQ) and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on digoxin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
liter per hour | 15.9 (21.5) | 13.4 (23.7)

27. Secondary Outcome: Part 1: Apparent Total Body Clearance From Plasma (CL/F) of Metformin
Description: CL/f was calculated as Dose/AUC0-inf, where AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. AUC0-inf was calculated as AUC0-tlast + Clast pred/Lambda Z, where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down); Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on metformin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
liter per hour | 495 (23.3) | 237 (77.1)

28. Secondary Outcome: Part 1: Apparent Total Body Clearance From Plasma (CL/F) of Rosuvastatin
Description: CL/f was calculated as Dose/AUC0-inf, where AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. AUC0-inf was calculated as AUC0-tlast + Clast pred/Lambda Z, where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down); Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on rosuvastatin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 11 | 11
liter per hour | 289 (64.3) | 292 (74.7)

29. Secondary Outcome: Part 2: Apparent Total Body Clearance From Plasma (CL/F) of Sumatriptan
Description: CL/f was calculated as Dose/AUC0-inf, where AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. AUC0-inf was calculated as AUC0-tlast + Clast pred/Lambda Z, where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down); Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on sumatriptan in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Part 2: Sumatriptan | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 19 | 19
liter per hour | 476 (43.7) | 533 (41.0)

30. Secondary Outcome: Part 1: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Digoxin
Description: Vz/f: the distribution of a study drug between plasma and the rest of the body after oral dosing. For single dose Vz/f = Dose/(AUC0-inf*Lambda Z), where AUC0-inf = (AUC0-tlast + Clast pred/Lambda Z), where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down); Clastpred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on digoxin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
liters | 787 (30.6) | 861 (34.5)

31. Secondary Outcome: Part 1: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Metformin
Description: Vz/f: the distribution of a study drug between plasma and the rest of the body after oral dosing. For single dose Vz/f = Dose/(AUC0-inf*Lambda Z), where AUC0-inf = (AUC0-tlast + Clast pred/Lambda Z), where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down); Clastpred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on metformin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
liters | 2206 (33.3) | 1389 (80.9)

32. Secondary Outcome: Part 1: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Rosuvastatin
Description: Vz/f: the distribution of a study drug between plasma and the rest of the body after oral dosing. For single dose Vz/f = Dose/(AUC0-inf*Lambda Z), where AUC0-inf = (AUC0-tlast + Clast pred/Lambda Z), where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down); Clastpred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and Lambda Z = the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on rosuvastatin in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 10
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 11 | 11
liters | 6712 (51.5) | 5789 (68.1)

33. Secondary Outcome: Part 2: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Sumatriptan
Description: Vz/f: the distribution of a study drug between plasma and the rest of the body after oral dosing. For single dose Vz/f = Dose/(AUC0-inf*Lambda Z), where AUC0-inf = (AUC0-tlast + Clast pred/Lambda Z), where AUC0-tlast was the AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down); Clastpred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and Lambda Z = the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on sumatriptan in this outcome measure.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Days 1 and 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 2: Sumatriptan | Part 2: Evobrutinib + Sumatriptan
Number analyzed (Participants) | 19 | 19
liters | 2193 (58.4) | 3007 (46.3)

34. Secondary Outcome: Part 1: Cumulative Amount Excreted (CAE) From Time Zero to the End of the Collection Interval After Dosing Dosing (Ae0-36) of Metformin
Description: Ae0-36 was calculated as the cumulative amount excreted from time zero (= dosing time) to the end of the collection interval after dosing, for metformin only. The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on metformin in this outcome measure.
Time Frame: Pre-dose, 0 to 4, 4 to 8, 8 to 12; 12 to 24 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams (mg)
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
milligrams (mg) | 0.574 (37.5) | 1.24 (62.3)

35. Secondary Outcome: Part 1: Renal Clearance (CLr) of Metformin
Description: CLr was calculated as Ae0-36 divided by AUC0-36, for metformin only. AUC0-36: AUC from time zero (= dosing time) to 36 hours post-dose (metformin only) calculated using the mixed log-linear trapezoidal rule (linear up, log down). The transporter cocktail included digoxin, metformin, and rosuvastatin. As pre-specified in protocol, data was analyzed and reported to characterize the effect of evobrutinib on metformin in this outcome measure.
Time Frame: Pre-dose, 0 to 4, 4 to 8, 8 to 12; 12 to 24 hours post-dose on Days 1 and 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib + Cocktail
Number analyzed (Participants) | 18 | 18
liter per hour | 28.5 (37.9) | 29.7 (26.1)

ADVERSE EVENTS:
Time Frame: Part 1: Cocktail Alone - Day 1 to Day 3; Evobrutinib Alone - Day 4 to Day 9; Evobrutinib + Cocktail - Day 10 to Day 12; Part 2: Sumatriptan Alone - Day 1; Evobrutinib Alone - Day 2 to Day 7; Evobrutinib + Sumatriptan - Day 8
Arm/Group | Part 1: Cocktail | Part 1: Evobrutinib | Part 1: Evobrutinib + Cocktail | Part 2: Sumatriptan | Part 2: Evobrutinib | Part 2: Evobrutinib + Sumatriptan
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 9/20 | 6/19 | 6/20 | 10/20 | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cocktail (N=20) | Part 1: Evobrutinib (N=20) | Part 1: Evobrutinib + Cocktail (N=19) | Part 2: Sumatriptan (N=20) | Part 2: Evobrutinib (N=20) | Part 2: Evobrutinib + Sumatriptan (N=20)
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 0 | 1 | 3 | 4 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT05064488/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT05064488/SAP_001.pdf